CLINICAL TRIAL: NCT03282617
Title: Dendritic Cell Therapy With CD137L-DC-EBV-VAX in Locally Advanced Stage IV or Locally Recurrent/Metastatic Nasopharyngeal Carcinoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NP01/03/16
Record Dates: First submitted 2017-09-12; First posted 2017-09-14 (Actual); Last update posted 2017-09-14 (Actual); Status verified 2017-09

CONDITIONS: Nasopharyngeal Cancer
MeSH Terms: conditions — Nasopharyngeal Neoplasms

STUDY DESIGN:
Intervention Model Description: Patients will be given CD137L-DC-EBV-VAX for about 5 - 7 times and be followed up until a maximum of 3 years from study entry.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- locally recurrent or metastatic nasopharyngeal cancer (Experimental): This cohort consists of patients with metastatic or locally recurrent NPC who have received systemic concurrent chemotherapy and have a favourable response of stable disease, partial or complete response. As up to 30% of these patients will suffer from relapse within 5 months of completion of chemotherapy, following definitive treatment, y, and treatment with CD137L-DC-EBV-VAX may activate T cell response against the tumor and prolong time to progression.
  Interventions: Biological: CD137L-DC-EBV-VAX
- stage 4 locally advanced nasopharyngeal cancer (Experimental): This cohort consists of patients with stage 4 locally advanced patients (N2 and N3 disease, and/or T4 disease) who are treated definitely with chemoradiation with curative intent, but who have a high risk of distant relapse. Treatment with CD137L-DC-EBV-VAX may activate antitumor T cell responses and prolong time to relapse.
  Interventions: Biological: CD137L-DC-EBV-VAX

INTERVENTIONS:
Biological: CD137L-DC-EBV-VAX — Patients will receive CD137L-DC-EBV-VAX at a dose of approximately 5-50 millioncells every 2 weeks, for a total of 5-7 times.
  Other Names: Dendritic cell therapy

SUMMARY:
This study is carried out to find out the safety and recommended dose of CD137L-DC-EBV-VAX in nasopharyngeal cancer. CD137L-DC-EBV-VAX is a product made from one of our own immune system cells (dendritic cell, DC). Dendritic cells are immune cells that help to stimulate our body's T lymphocytes to fight cancer by presenting specific proteins from the cancer cells. The investigators have developed in the laboratory a highly effective dendritic cell which is primed to activate T cells with the Epstein-Barr virus (EBV) proteins. It is hoped that this will stir an immune response to recognize NPC cells and kill them as part of body's immune surveillance system.

DETAILED DESCRIPTION:
This study will involve two cohorts of patients, A and B. Patients are invited because they have either (A) locally recurrent or metastatic nasopharyngeal cancer; or (B) stage 4 locally advanced nasopharyngeal cancer (N2 or N3 disease and/or T4) and is known to be associated with a high risk of distant relapse.

This study is carried out to find out the safety and recommended dose of CD137L-DC-EBV-VAX in nasopharyngeal cancer. CD137L-DC-EBV-VAX is a product made from one of our own immune system cells (dendritic cell, DC). Dendritic cells are immune cells that help to stimulate our body's T lymphocytes to fight cancer by presenting specific proteins from the cancer cells. The investigators have developed in the laboratory a highly effective dendritic cell which is primed to activate T cells with the Epstein-Barr virus (EBV) proteins. It is hoped that this will stir an immune response to recognize NPC cells and kill them as part of body's immune surveillance system.

ELIGIBILITY:
Eligibility Criteria:

* Age ≥ 18 year
* Ability to understand and the willingness to sign a written informed consent document.
* 2 cohorts of patients are eligible for the study: Cohort A - Histologically or cytologically confirmed non-keratinizing nasopharyngeal carcinoma (NPC) that has recurred at locoregional and/or distant sites. Patients must have just received at least 1 cycle of chemotherapy and achieved stable disease, partial or complete response.

Cohort B - Histologically or cytologically confirmed stage 4A/B (locally advanced) non-keratinizing NPC that has just completed concurrent chemoradiotherapy less than 2 months before study entry.

* Measurable disease according to the RECIST criteria (version 1.1) is not necessary, but tumor assessments on follow up will be according to RECIST criteria (version 1.1) as defined in section 11 for the evaluation of disease.
* Archived or fresh tumor sample available. Willingness to donate blood and tissue for mandatory correlative research studies (see Section 9).
* ECOG performance status of 0, 1 or 2 (see Appendix A).
* Patients must have adequate organ and marrow function as defined below:

  * Absolute monocyte count ≥0.2 x 109/L
  * Platelets ≥100 x109/L
  * Hemoglobin ≥8.0 g/dL
  * Serum alanine aminotransferase (ALT; serum glutamate-pyruvate transferase, [SGPT]) < 2.5 x upper limit of normal (ULN), OR < 5 x ULN in the presence of liver metastases.
  * Serum total bilirubin < 2 x ULN (except patients with Gilbert Syndrome, who can have total bilirubin <3.0 mg/dL)
  * Serum creatinine < 1.5 x ULN

Exclusion Criteria:

- Any of the following:

* Chemotherapy ≤ 4 weeks prior to CD137L-DC-EBV-VAX study treatment.
* Radiotherapy ≤ 4 weeks prior to CD137L-DC-EBV-VAX study treatment.
* Nitrosoureas or Mitomycin C ≤ 4 weeks prior to registration

NOTE: Prior palliative radiotherapy to bone metastases is allowed ≤ 4 weeks prior to registration. Prior immunotherapy with immune checkpoint inhibitors will not be allowed.

* Prior investigational agents ≤ 4 weeks prior to registration.
* Known allergy to Tetanus and/or Diphtheria toxoid.
* Known brain metastases or leptomeningeal metastases. NOTE: symptomatic, and/or if they require immunosuppressive doses of corticosteroids (e.g. >10 mg/day prednisone or equivalents) for at least 2 weeks prior to study drug administration. Patients with treated brain metastases who are deemed clinically stable and without radiological progression on PET, MRI or CT scan performed ≤ 8 weeks of study entry, are not excluded. NOTE: Primary nasopharyngeal cancers that directly invade the skull base and extend into the infratemporal fossa(e) are not regarded as brain metastases and are not excluded.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Any of the following:

  * Pregnant women
  * Nursing women
  * Men or women of childbearing potential who are unwilling to employ adequate contraception
* Active autoimmune disease or history of autoimmune disease that might recur, which may affect vital organ function or require immune suppressive treatment including systemic corticosteroids. NOTE: These include but are not limited to patients with a history of immune related neurologic disease, multiple sclerosis, autoimmune (demyelinating) neuropathy, Guillain-Barre syndrome, myasthenia gravis; systemic autoimmune disease such as SLE, connective tissue diseases, scleroderma, inflammatory bowel disease (IBD), Crohn's, ulcerative colitis, hepatitis; and patients with a history of toxic epidermal necrolysis (TEN), Stevens-Johnson syndrome, or phospholipid syndrome should be excluded because of the risk of recurrence or exacerbation of disease. Patients with vitiligo, endocrine deficiencies including thyroiditis managed with replacement hormones including physiologic corticosteroids are eligible. Patients with rheumatoid arthritis and other arthropathies, Sjögren's syndrome and psoriasis controlled with topical medication and patients with positive serology, such as antinuclear antibodies (ANA), anti-thyroid antibodies should be evaluated for the presence of target organ involvement and potential need for systemic treatment but should otherwise be eligible.
* Patients are permitted to enroll if they have vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger (precipitating event).
* Condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses <10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease. Patients are permitted to use topical, ocular, intra-articular, intranasal, and inhalational corticosteroids (with minimal systemic absorption). Physiologic replacement doses of systemic corticosteroids are permitted, even if <10 mg/day prednisone equivalents. A brief course of corticosteroids for prophylaxis (e.g., contrast dye allergy) or for treatment of non-autoimmune conditions (e.g., delayed-type hypersensitivity reaction caused by contact allergen) is permitted.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2017-08-14 (Actual); Primary Completion 2019-08-14 (Estimated); Study Completion 2020-08-14 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability and recommended dose of CD137L-DC-EBV-VAX | From the start of assessment until study completion, an average of 3 year

SECONDARY OUTCOMES:
Activation of EBV-specific T cell responses | From the start of assessment until study completion, an average of 3 year
Antitumor Effect based on Immune Response Criteria (IRC) | From the start of assessment until study completion, an average of 3 year
Progression-free survival and overall survival | From the start of assessment until study completion, an average of 3 year

CONTACTS AND LOCATIONS:
Overall Officials: Boon Cher Goh, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Petersson F. Nasopharyngeal carcinoma: a review. Semin Diagn Pathol. 2015 Jan;32(1):54-73. doi: 10.1053/j.semdp.2015.02.021. Epub 2015 Feb 25. PMID 25769204
- [Background] Lee AW, Ma BB, Ng WT, Chan AT. Management of Nasopharyngeal Carcinoma: Current Practice and Future Perspective. J Clin Oncol. 2015 Oct 10;33(29):3356-64. doi: 10.1200/JCO.2015.60.9347. Epub 2015 Sep 8. PMID 26351355
- [Background] Yu MC, Yuan JM. Epidemiology of nasopharyngeal carcinoma. Semin Cancer Biol. 2002 Dec;12(6):421-9. doi: 10.1016/s1044579x02000858. PMID 12450728